CLINICAL TRIAL: NCT01113177
Title: Effect of Functional Treatment on Mandibular Asymmetry Caused by Unilateral Temporomandibular Joint Involvement in Children With Juvenile Idiopathic Arthritis
Brief Title: Effect of Functional Treatment on Mandibular Asymmetric Growth
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Thomas Klit Pedersen, Dep. of orthodontics
Other Study IDs: AU-2010
Record Dates: First submitted 2010-03-15; First posted 2010-04-29 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Temporomandibular Joint Disorder
Keywords: Mandibular growth temporomandibular arthritis
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Distraction splint therapy: All JIA patients with asymmetric mandibular growth due to unilateral TMJ arthritis are offered non-surgical functional orthodontic splint therapy with a distraction splint. Mandibular growth is thereafter evaluated in the affected side compared with the mandibular growth in the healthy side of the same individual.
  Interventions: Device: Distraction splint therapy

INTERVENTIONS:
Device: Distraction splint therapy — After the diagnosis of unilateral TMJ arthritis with clinical asymmetric mandibular growth deviations the JIA patients are offered treatment with a distraction splint. The appliance consists of an acrylic splint (distraction splint) covering the occlusal surfaces of the teeth in the upper or lower dental arch. The height of the splint is thereafter gradually increased every 6th to 10th weeks in order to optimize the mandible growth in the affected side and thereby reduce the overall asymmetric mandibular growth pattern(non-surgical distraction of the TMJ and mandibular condyle).
  Other Names: functional appliance

SUMMARY:
Temporomandibular joint (TMJ) arthritis is known to alter the mandibular development in children diagnosed with juvenile idiopathic arthritis. In a number of cases a genuine breakdown of cartilage and bone is seen in the affected joint which leads to asymmetric mandibular growth in the affected side. In cases of unilateral TMJ involvements severe mandibular asymmetric mandibular growth deviations are seen. We hypothesize that these growth deviations can be minimized and controlled by the use functional orthodontic appliance therapy.

DETAILED DESCRIPTION:
This is a retrospective study design with the aim to evaluate the clinical procedures we have used the last 15 years to treat JIA patients with unilateral TMJ arthritis. More specifically, the purpose is to evaluate the mandibular growth in all JIA patients with unilateral TMJ arthritis and an asymmetric mandibular growth pattern treated with non-surgical distraction splint therapy between 1994 and 2010 at the dep. of Orthodontics, Aarhus University, Denmark. The evaluation is based on radiological examinations at the beginning of their non-surgical distraction treatment as well as after the patients have finished their distraction-splint therapy.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile Idiopathic arthritis patients diagnosed with unilateral temporomandibular joint arthritis and an asymmetric mandibular growth pattern

Exclusion Criteria:

* Juvenile Idiopathic arthritis patients diagnosed with bilateral temporomandibular joint arthritis
* Juvenile Idiopathic arthritis patients with no mandibular growth potential left.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Juvenile Idiopathic arthritis patients diagnosed with unilateral temporomandibular joint arthritis and an asymmetric mandibular growth pattern
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 1994-06; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Mandibular growth in children with unilateral TMJ arthritis treated with an acrylic distraction splint | average treatment with splint is 6.4 years
  The craniofacial dimensions are measured radiologically prior to the start of the treatment with the distraction splint. Second measurements of the craniofacial dimensions are evaluated after the patients have ended the treatment with the distraction splint. In that way we are able to evaluate the craniofacial growth in the affected side compared to the craniofacial growth in the "healthy" side in JIA patients with unilateral TMJ arthritis. The succces of the distraction splint treatment is decided based the splints ability to normalize the craniofacial growth in the affacted side.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Pedersen, DDS Ph.D, Study Director
Locations (1):
- Dep. of Orthodontics, Aarhus University, Aarhus, Denmark